CLINICAL TRIAL: NCT04083235
Title: An Open-label, Randomised, Multicentre, Phase III Study of Irinotecan Liposome Injection, Oxaliplatin, 5-fluorouracil/Leucovorin Versus Nab-paclitaxel Plus Gemcitabine in Subjects Who Have Not Previously Received Chemotherapy for Metastatic Adenocarcinoma of the Pancreas
Brief Title: A Study to Assess the Effectiveness and Safety of Irinotecan Liposome Injection, 5-fluorouracil/Leucovorin Plus Oxaliplatin in Patients Not Previously Treated for Metastatic Pancreatic Cancer, Compared to Nab-paclitaxel+Gemcitabine Treatment
Acronym: NAPOLI 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-US-60010-001; 2018-003585-14 (EudraCT Number)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Adenocarcinoma of the Pancreas
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Irinotecan liposome injection + Oxaliplatin + 5-FU/LV (Experimental): Irinotecan liposome injection, oxaliplatin, 5 FU/LV, will be administered on Days 1 and 15 of each 28-day cycle (until progression or unacceptable toxicity).
  Interventions: Drug: Irinotecan Liposomal Injection; Drug: Oxaliplatin; Drug: 5Fluorouracil; Drug: Leucovorin
- Nab-paclitaxel + Gemcitabine (Active Comparator): Nab-paclitaxel and gemcitabine will be administered on Days 1, 8 and 15 of each 28-day cycle (until progression or unacceptable toxicity).
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Irinotecan Liposomal Injection — Irinotecan liposome injection is irinotecan in the form of the sucrosofate salt, encapsulated in liposomes for i.v. infusion. It is supplied in sterile, single-use vials containing 10 mL of irinotecan liposome injection at a concentration of 4.3 mg/mL free base equivalent (FBE).
  Other Names: Onivyde®; Nal-IRI
  Arms: Irinotecan liposome injection + Oxaliplatin + 5-FU/LV
Drug: Oxaliplatin — Oxaliplatin injection, USP is supplied in single-dose vials containing 50 mg, 100 mg or 200 mg of oxaliplatin as a sterile, preservative-free, aqueous solution at a concentration of 5 mg/mL.
  Other Names: Eloxatin®
  Arms: Irinotecan liposome injection + Oxaliplatin + 5-FU/LV
Drug: 5Fluorouracil — Fluorouracil injection, USP is a colorless to faint yellow, aqueous, sterile, nonpyrogenic injectable solution available in 50 mL and 100 mL pharmacy bulk package. Each mL contains 50 mg fluorouracil in water for injection, USP.
  Other Names: Adrucil®; flurouracil; 5-FU
  Arms: Irinotecan liposome injection + Oxaliplatin + 5-FU/LV
Drug: Leucovorin — Leucovorin Calcium for Injection is supplied in vials ranging from 50-500 mg and available as an injectable solution or lyophilized powder for reconstitution.
  Other Names: Folinic Acid
  Arms: Irinotecan liposome injection + Oxaliplatin + 5-FU/LV
Drug: Nab-paclitaxel — Nab-paclitaxel is a lyophilised powder containing 100 or 250 mg of paclitaxel formulated as albumin-bound particles in single-use vials for re-constitution. Each mL of the reconstituted formulation will contain 5 mg/mL paclitaxel.
  Other Names: Abraxane®
  Arms: Nab-paclitaxel + Gemcitabine
Drug: Gemcitabine — Gemcitabine for injection is a lyophilised powder for solution for infusion, with each single use vial containing 200 mg, 1 g or 2 g of gemcitabine.
  Other Names: Gemzar®
  Arms: Nab-paclitaxel + Gemcitabine

SUMMARY:
The purpose of this study is to look at the efficacy and safety of Irinotecan liposome injection in combination with other approved drugs used for cancer therapy, namely 5 fluorouracil/leucovorin (5FU/LV) plus oxaliplatin compared to nab-paclitaxel + gemcitabine treatment in improving the overall survival of patients not previously treated for metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytologically confirmed adenocarcinoma of the pancreas that has not been previously treated in the metastatic setting.
* Initial diagnosis of metastatic disease must have occurred ≤6 weeks prior to screening.
* Subject has one or more metastatic lesions measurable by computed tomography (CT) scan (or magnetic resonance imaging (MRI), if the subject is allergic to CT contrast media) according to RECIST Version 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject has adequate biological parameters as demonstrated by the following blood counts:(a) Absolute neutrophil count (ANC) ≥2000/mm3 without the use of hemopoietic growth factors within the last 7 days prior to randomisation (b) Platelet count ≥100,000/mm3 (c) Haemoglobin (Hgb) ≥9 g/dL obtained ≤14 days prior to randomisation.
* Adequate hepatic function as evidenced by: (a) Serum total bilirubin ≤1.5x ULN (biliary drainage is allowed for biliary obstruction), and (b) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5x upper limit of normal (ULN) (≤5x ULN is acceptable if liver metastases are present).
* Adequate renal function as evidenced by creatinine clearance ≥30 mL/min.
* Adequate coagulation studies (obtained ≤14 days prior to randomisation) as demonstrated by prothrombin time and partial thromboplastin time within normal limits (≤1.5xULN ).

Exclusion Criteria:

* Prior treatment of pancreatic cancer in the metastatic setting with surgery, radiotherapy, chemotherapy or investigational therapy
* Prior treatment of pancreatic adenocarcinoma with chemotherapy in the adjuvant setting, except those where at least 12 months have elapsed since completion of the last dose and no persistent treatment-related toxicities are present.
* Subject has only localised advanced disease.
* Documented serum albumin <3 g/dL
* Known history of central nervous system (CNS) metastases.
* Clinically significant gastrointestinal disorder
* History of any second malignancy in the last 2 years
* Concurrent illnesses that would be a relative contraindication to trial participation
* Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1
* Neuroendocrine (carcinoid, islet cell) or acinar pancreatic carcinoma
* Known low or absent dihydropyrimidine dehydrogenase (DPD) activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2025-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (199):
- United States (72):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Health- MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic - Scottsdale, Phoenix, Arizona
  - Comprehensive Blood And Cancer Center, Bakersfield, California
  - University of California- Irvine Health Cancer Cente, Costa Mesa, California
  - City of Hope National Medical Center, Duarte, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - St. Jude Hospital Yorba Linda dba St. Joseph Heritage Healthcare, Orange, California
  - University of California - Irvine Medical Center, Orange, California
  - Torrance Memorial Physician Network Cancer Care, Redondo Beach, California
  - Sutter Health Sacramento, Sacramento, California
  - Presbyterian Intercommunity Hospital (PIH), Whittier, California
  - UC Health Memorial Hospital, Colorado Springs, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center of Florida, Inc., Miami Beach, Florida
  - Florida Cancer Specialists - Fort Myers, Sarasota, Florida
  - Florida Cancer Specialists - Panhandle, Tallahassee, Florida
  - Florida Cancer Specialists - St. Petersburg, Tampa, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Edward Hospital - Elmhurst, Elmhurst, Illinois
  - Illinois CancerCare - Peoria, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Siouxland Hematology - Oncology Associates, LLP, Sioux City, Iowa
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Beth Israel Deaconess, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Health Partners Institute, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Research Medical Center, Kansas City, Missouri
  - Frontier Cancer Center, Billings, Montana
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Clinical Research Alliance, Inc, Lake Success, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Messino Cancer Center, Asheville, North Carolina
  - The Ohio State University Comprehensive Cancer Center - Arthur G. James Cancer Hospital and Richard J. Solovev Research Institute (OSUCCC - James), Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - University of Oklahoma - Health Sciences Center, Oklahoma City, Oklahoma
  - Oncology Associates of Oregon, Eugene, Oregon
  - Compass Oncology - Rose Quarter Cancer Center, Portland, Oregon
  - Kaiser Permanente - Northwest, Portland, Oregon
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Chattanooga Oncology Hematology Care - Tennessee Oncology, Chattanooga, Tennessee
  - The West Cancer Center, Memphis, Tennessee
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology - Wichita Falls, Wichita Falls, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Blue Ridge Cancer Care, Wytheville, Virginia
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Bankstown-Lidcombe Hospital, Bankstown
  - Monash Medical Centre, Clayton
  - Fiona Stanley Hospital, Murdoch
  - Sir Charles Gairdner Hospital, Nedlands
  - St John of God Subiaco Hospital, Subiaco
  - Queen Elizabeth Hospital, Woodville South
- Austria (4):
  - Medizinische Universitaet Graz, Graz
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - SCRI-CCCIT Gemeinnutzige Gmbh- Gemeinnutzige Salzburger Landeskliniken Betriebsgesmbh, Salzburg
  - Medical University of Vienna, Vienna
- Belgium (7):
  - Onze-Lieve-Vrouwziekenhuis, Aalst
  - ASBL Grand Hôpital de Charleroi (GHdC), Site Notre Dame, Charleroi
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
  - University Hospital Gent, Ghent
  - Hospital centre Jolimont, Haine-Saint-Paul
  - University Hospital (UZ) Leuven, Leuven
  - University Hospital Mont-Godinne, Yvoir
- Brazil (15):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - Centro Regional Integrado de Oncologia (CRIO), Ceará
  - Instituto de Oncologia do Parana - IOP, Curitiba
  - Centro de Pesquisas Oncológicas - CEPON, Florianópolis
  - Hospital de Caridade de Ijui, Ijuí
  - Clinica Neoplasias Litoral, Itajaí
  - Hospital Bruno Born, Lajeado
  - Centro de Pesquisas Clinicas de Natal - CPCLIN, Natal
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Instituto Nacional Do Cancer (INCA), Rio de Janeiro
  - Instituto COI, Rio de Janeiro
  - CIP Centro Integrado de Pesquisas do Hospital de Base, São José do Rio Preto
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Instituto Brasileiro de Controle do Cancer - IBCC (Sao Paulo), São Paulo
  - Instituto do Cancer do Estado de São Paulo (ICESP), São Paulo
- Canada (4):
  - Alberta Health Services Cross Cancer Institute, Edmonton
  - Queen Elizabeth II Health Sciences Centre, Halifax
  - McGill University Faculty of Medicine - Royal Victoria Hospital, Montreal
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Department of Oncology, Olomouc
  - Thomayerova Nemocnice, Prague
- France (10):
  - CHRU de Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Centre Oscar Lambret, Lille
  - Hôpital Edouard Herriot, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Centre Antoine-Lacassagne, Nice
  - Hopital Saint Louis, Paris
  - CHU Bordeaux - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Universitaire de Poitiers - Poitiers University Hospital, Poitiers
  - Strasbourg Oncologie Liberale, Strasbourg
- Germany (15):
  - Charité - Universitaetsmedizin Berlin, Berlin
  - St. Josef-Hospital, Bochum
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Krankenhaus Nordwest, Frankfurt
  - Studiengesellschaft BSF, Halle
  - Martin Luther Universitat Halle-Wittenberg, Halle
  - Facharztzentrum Eppendorf, Hamburg
  - Marienkrankenhaus Hamburg, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Slk-Kliniken, Heilbronn
  - Klinikum Mannheim, Mannheim
  - Krankenhaus St. Franziskus - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
- Greece (5):
  - Agios Savvas Anticancer Hospital, Athens
  - General Hospital of Athens - Laiko, Athens
  - National and Kapodistrian University of Athens, Athens
  - University General Hospital of Ioannina, Ioannina
  - Theagenion Hospital, Thessaloniki
- Hungary (6):
  - Dél-pesti Centrumkórház - Szent László Kórház telephely, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Semmelweis Egyetem Belgyógyászati és Hematológiai Klinika, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelointézet, Szolnok
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
- Italy (8):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - AUSL di Piacenza-Ospedale Guglielmo Da Saliceto, Piacenza
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - AOU Ospedali Riuniti di Ancona, Torrette
  - Azienda Ospedaliera - Universitaria Integrata di Verona - Ospedale Borgo Roma, Verona
- Portugal (5):
  - Hospital de Braga, Braga
  - Champalimaud Cancer Center, Lisbon
  - Centro Hospitalar Universitario de Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude Matosinhos E.P.E. Hospital Pedro Hispano, Senhora da Hora
  - Centro Hospitalar de Vila Nova de Gaia/Espinho EPE, Vila Nova de Gaia
- Russia (6):
  - Evimed LLC, Chelyabinsk
  - Limited Liability Company- Clinica Druzhkovyh, Kazan'
  - Kursk Regional Clinical Oncology Dispensary, Kursk
  - Main Military Clinical Hospital named after N.N. Burdenko, Moscow
  - Federal State Budgetary Institution - Russian Scientific Center of Radiology and Surgical Technologies n.a. academician A.M.Granov, Saint Petersburg
  - Volga District Medical Centre, Veliky Novgorod
- South Korea (6):
  - Inje University Haeundae Paik Hospital, Busan
  - National Cancer Center, Goyang-si
  - CHA Bundang Medical Center, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (19):
  - Hospital General Universitario de Elche, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau Barcelona, Barcelona
  - Hospital Vall D Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Corporacio Sanitaria Parc Tauli - Hospital de Sabadell, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Complejo Hospitalario Universitario de Granada - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (5):
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - Royal Marsden Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Cancer Research UK - Christie Hospital Foundation NHS Trust - Dept of Medical Oncology, Manchester
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Wainberg ZA, Melisi D, Macarulla T, Pazo Cid R, Chandana SR, De La Fouchardiere C, Dean A, Kiss I, Lee WJ, Goetze TO, Van Cutsem E, Paulson AS, Bekaii-Saab T, Pant S, Hubner RA, Xiao Z, Chen H, Benzaghou F, O'Reilly EM. NALIRIFOX versus nab-paclitaxel and gemcitabine in treatment-naive patients with metastatic pancreatic ductal adenocarcinoma (NAPOLI 3): a randomised, open-label, phase 3 trial. Lancet. 2023 Oct 7;402(10409):1272-1281. doi: 10.1016/S0140-6736(23)01366-1. Epub 2023 Sep 11. PMID 37708904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, open-label study was conducted in participants with metastatic adenocarcinoma of the pancreas at 187 investigational sites in 18 countries (Australia, Brazil, Canada, Israel, Republic of Korea, United States, Austria, Belgium, Czechia, France, Germany, Greece, Hungary, Italy, Portugal, Spain, United Kingdom, and Russia). First participant was recruited on 11 February 2020 and data cut-off (DCO) date was 23 July 2022.
Pre-assignment Details: This study consisted of a screening period (up to 28 days), treatment period (28-day cycles of treatment until radiologically determined disease progression per response evaluation criteria in solid tumors [RECIST 1.1]), unacceptable study medication related toxicity or withdrawal from study treatment followed by survival follow-up (until death or study closure, whichever occurred first). A total of 770 participants were randomized in 1:1 ratio using an interactive web response system (IWRS).
Groups:
- NALIRIFOX: Participants were treated with irinotecan liposome injection 50 milligram per square meter (mg/m^2) followed by oxaliplatin 60 mg/m^2, followed by leucovorin (LV) 400 mg/m^2 and then 5-fluorouracil (FU) 2400 mg/m^2 intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Nab-paclitaxel+Gemcitabine: Participants were treated with nab-paclitaxel 125 mg/m^2 followed by gemcitabine 1000 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | NALIRIFOX | Nab-paclitaxel+Gemcitabine
Started | 383 | 387
Received Treatment | 370 | 379
Completed | 59 | 77
Not Completed | 324 | 310
Not completed — Death | 252 | 277
Not completed — Withdrawal by Subject | 13 | 17
Not completed — Lost to Follow-up | 1 | 1
Not completed — Does not meet entry criteria | 1 | 0
Not completed — Did not receive treatment | 13 | 8
Not completed — Ongoing at the time of DCO | 44 | 7

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population consisted of all randomized participants to whom study treatment was assigned by randomization.
Groups:
- NALIRIFOX: Participants were treated with irinotecan liposome injection 50 mg/m^2 followed by oxaliplatin 60 mg/m^2, followed by LV 400 mg/m^2 and then 5-FU 2400 mg/m^2 IV infusion on Days 1 and 15 of each 28-day cycle until disease progression, death, unacceptable study treatment-related toxicity or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | NALIRIFOX | Nab-paclitaxel+Gemcitabine | Total
Number analyzed (Participants) | 383 | 387 | 770
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.71) | 64.0 (8.34) | 63.4 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 157 | 336
  Male | 204 | 230 | 434
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 30 | 79
  Not Hispanic or Latino | 305 | 328 | 633
  Unknown or Not Reported | 29 | 29 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 315 | 324 | 639
  Not Reported | 26 | 29 | 55
  Asian | 20 | 18 | 38
  Black or African American | 12 | 7 | 19
  Other | 7 | 6 | 13
  Multiple | 3 | 0 | 3
  American Indian or Alaska Native | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The OS was defined as time from the date of randomization to the date of death due to any cause. Participants who did not have a date of death recorded at the time of the final analysis were censored at the last known time that the participant was alive. The median OS was measured using Kaplan-Meier technique.
Time Frame: Assessments performed at baseline (within 28 days before start of study treatment), every 8 weeks after first dose, end of treatment (EoT) visit, then every 2 months thereafter up to DCO date of 23 July 2022 (maximum of 893 days)
Population: The ITT population consisted of all randomized participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NALIRIFOX | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 383 | 387
months | 11.1 [10.0 to 12.1] | 9.2 [8.3 to 10.6]
Statistical Analysis 1: Comparison: NALIRIFOX vs Nab-paclitaxel+Gemcitabine; Test type: Other; p = 0.04, Stratified log-rank test; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.70 to 0.99] — The HR and 95% confidence interval (CI) was based on a stratified Cox proportional hazards regression model, stratified by baseline Eastern Cooperative Oncology Group (ECOG) performance status, region and liver metastases as per IWRS

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the first documented disease progression using response evaluation criteria in solid tumors (RECIST) Version 1.1 as per Investigator assessment or death due to any cause. The median PFS was measured using Kaplan-Meier technique.
Time Frame: Assessments performed at baseline (within 28 days before start of study treatment), every 8 weeks after first dose until EoT visit (maximum of 893 days)
Population: The ITT population consisted of all randomized participants to whom study treatment was assigned by randomization. Only participants with PFS event are reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NALIRIFOX | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 249 | 259
months | 7.4 [6.0 to 7.7] | 5.6 [5.3 to 5.8]
Statistical Analysis 1: Comparison: NALIRIFOX vs Nab-paclitaxel+Gemcitabine; Test type: Other; p < 0.0001, Stratified log-rank test; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.58 to 0.83] — The HR and 95% CI was based on a stratified Cox proportional hazards regression model, stratified by baseline ECOG performance status, region and liver metastases as per IWRS

3. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with a best overall response (BOR) characterized as either a complete response (CR) or partial response (PR) per RECIST Version 1.1. BOR was defined as the best response as recorded from randomization until documented objective disease progression using RECIST Version 1.1. As per RECIST version 1.1, CR is disappearance of all target lesions; PR is >=30% decrease in the sum of the longest diameter of target lesions; and overall response = CR + PR. The ORR was calculated using Clopper-Pearson method.
Time Frame: Assessments performed at baseline (within 28 days before start of study treatment), every 8 weeks after first dose until EoT visit, (maximum of 893 days)
Population: The ITT population consisted of all randomized participants to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NALIRIFOX | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 383 | 387
percentage of participants | 41.8 [36.8 to 46.9] | 36.2 [31.4 to 41.2]
Statistical Analysis 1: Comparison: NALIRIFOX vs Nab-paclitaxel+Gemcitabine; Test type: Other; p = 0.11, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.95 to 1.69] — OR, 95% CI and p-value were obtained from the Cochran-Mantel-Haenszel test adjusting by baseline ECOG performance status, region and liver metastases as per IWRS

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported from the time of first study treatment administration (Day 1) up to DCO date of 23 July 2022 (maximum of 893 days)
Description: The Safety population was a subset of the ITT population that received at least 1 dose (including a partial dose) of any component of the study medication in the combination.
Arm/Group | NALIRIFOX | Nab-paclitaxel+Gemcitabine
All-Cause Mortality (participants affected / at risk) | 252/370 | 277/379
Serious Adverse Events (participants affected / at risk) | 201/370 | 195/379
Other Adverse Events (participants affected / at risk) | 364/370 | 371/379
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NALIRIFOX (N=370) | Nab-paclitaxel+Gemcitabine (N=379)
Diarrhoea (Gastrointestinal disorders) | 23 (28) | 9 (9)
Vomiting (Gastrointestinal disorders) | 22 (26) | 6 (6)
Nausea (Gastrointestinal disorders) | 18 (24) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 8 (8)
COVID-19 (Infections and infestations) | 18 (18) | 14 (14)
Pneumonia (Infections and infestations) | 7 (7) | 13 (13)
Pyrexia (General disorders) | 8 (9) | 12 (14)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 8 (8)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 8 (8)
Ascites (Gastrointestinal disorders) | 6 (7) | 5 (6)
Colitis (Gastrointestinal disorders) | 7 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 6 (6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5) | 4 (4)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2)
Ileus (Gastrointestinal disorders) | 3 (3) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Duodenal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Terminal ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 16 (18)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
Biliary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3)
Febrile infection (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cholangitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder abscess (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Implant site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infective spondylitis (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Asthenia (General disorders) | 7 (7) | 2 (2)
Fatigue (General disorders) | 7 (7) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 6 (6)
Malaise (General disorders) | 3 (4) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Catheter site inflammation (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Inadequate analgesia (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 10 (11) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (9) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Embolism (Vascular disorders) | 1 (1) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Iliac vein occlusion (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 4 (4) | 6 (6)
Biliary obstruction (Hepatobiliary disorders) | 6 (6) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Pineal gland cyst (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (5) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 9 (10)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Penile vein thrombosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Priapism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NALIRIFOX (N=370) | Nab-paclitaxel+Gemcitabine (N=379)
Diarrhoea (Gastrointestinal disorders) | 258 (566) | 135 (221)
Nausea (Gastrointestinal disorders) | 215 (406) | 162 (216)
Vomiting (Gastrointestinal disorders) | 139 (222) | 96 (168)
Stomatitis (Gastrointestinal disorders) | 50 (81) | 45 (54)
Constipation (Gastrointestinal disorders) | 93 (115) | 113 (141)
Abdominal pain (Gastrointestinal disorders) | 92 (110) | 75 (80)
Dry mouth (Gastrointestinal disorders) | 28 (29) | 14 (16)
Fatigue (General disorders) | 120 (173) | 143 (183)
Asthenia (General disorders) | 110 (164) | 101 (166)
Oedema peripheral (General disorders) | 52 (60) | 107 (134)
Mucosal inflammation (General disorders) | 50 (60) | 16 (20)
Pyrexia (General disorders) | 33 (43) | 84 (129)
Neuropathy peripheral (Nervous system disorders) | 66 (89) | 66 (92)
Dysgeusia (Nervous system disorders) | 63 (74) | 58 (67)
Peripheral sensory neuropathy (Nervous system disorders) | 56 (79) | 51 (60)
Paraesthesia (Nervous system disorders) | 44 (53) | 33 (41)
Neutropenia (Blood and lymphatic system disorders) | 108 (264) | 121 (278)
Anaemia (Blood and lymphatic system disorders) | 94 (134) | 151 (196)
Thrombocytopenia (Blood and lymphatic system disorders) | 50 (93) | 84 (173)
Leukopenia (Blood and lymphatic system disorders) | 18 (40) | 24 (43)
Neutrophil count decreased (Investigations) | 73 (208) | 69 (126)
Platelet count decreased (Investigations) | 39 (71) | 67 (109)
Weight decreased (Investigations) | 82 (92) | 33 (34)
Alanine aminotransferase increased (Investigations) | 45 (64) | 48 (64)
Aspartate aminotransferase increased (Investigations) | 40 (58) | 40 (55)
White blood cell count decreased (Investigations) | 16 (24) | 32 (54)
Decreased appetite (Metabolism and nutrition disorders) | 132 (157) | 68 (136)
Hypokalaemia (Metabolism and nutrition disorders) | 116 (190) | 49 (70)
Dehydration (Metabolism and nutrition disorders) | 35 (40) | 29 (31)
Alopecia (Skin and subcutaneous tissue disorders) | 52 (53) | 119 (120)
Rash (Skin and subcutaneous tissue disorders) | 11 (12) | 34 (37)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 25 (30)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 43 (49)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 31 (43)
Abdominal pain upper (Gastrointestinal disorders) | 27 (34) | 21 (29)
Flatulence (Gastrointestinal disorders) | 30 (33) | 18 (21)
Dyspepsia (Gastrointestinal disorders) | 23 (32) | 18 (20)
Abdominal distension (Gastrointestinal disorders) | 22 (26) | 13 (15)
Haemorrhoids (Gastrointestinal disorders) | 19 (22) | 12 (13)
Chills (General disorders) | 6 (6) | 19 (20)
Dizziness (Nervous system disorders) | 24 (25) | 40 (44)
Headache (Nervous system disorders) | 23 (37) | 19 (24)
Polyneuropathy (Nervous system disorders) | 16 (19) | 19 (20)
Neurotoxicity (Nervous system disorders) | 21 (35) | 13 (22)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 26 (33) | 30 (31)
Hypomagnesaemia (Metabolism and nutrition disorders) | 34 (44) | 16 (22)
Hyponatraemia (Metabolism and nutrition disorders) | 18 (21) | 20 (21)
Gamma-glutamyltransferase increased (Investigations) | 44 (54) | 34 (35)
Blood alkaline phosphatase increased (Investigations) | 39 (42) | 31 (33)
Blood bilirubin increased (Investigations) | 21 (23) | 22 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (14) | 22 (26)
Urinary tract infection (Infections and infestations) | 27 (29) | 23 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (28) | 45 (48)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 24 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 30 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (37) | 33 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (16) | 30 (41)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 17 (22) | 21 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 30 (35)
Hypotension (Vascular disorders) | 21 (27) | 25 (26)
Hypertension (Vascular disorders) | 21 (24) | 15 (19)
Insomnia (Psychiatric disorders) | 28 (28) | 32 (32)
Anxiety (Psychiatric disorders) | 10 (10) | 24 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT04083235/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT04083235/SAP_001.pdf